CLINICAL TRIAL: NCT07100587
Title: The Effect of a Ketogenic vs. Mediterranean Diet on Metabolic and Hormonal Parameters in Patients With Active Acromegaly: A Prospective Crossover Study
Brief Title: Ketogenic vs. Mediterranean Diet on Metabolic and Hormonal Parameters in Patients With Active Acromegaly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Valentina Guarnotta, Professor, University of Palermo
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14
Record Dates: First submitted 2025-07-14; First posted 2025-08-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Acromegaly
Keywords: ketogenic diet; mediterranean diet
MeSH Terms: conditions — Acromegaly | interventions — Diet, Ketogenic; Diet, Mediterranean

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Ketogenic Diet (3 weeks) (Experimental): Participants will follow a structured ketogenic diet for 3 weeks (~1200 kcal/day, <30 g/day carbohydrates) to induce nutritional ketosis.
  Interventions: Behavioral: Ketogenic diet
- Arm B: Mediterranean Diet (Active Comparator): Following a 2-week transition phase, participants will switch to a Mediterranean diet for 3 weeks (~1200 kcal/day), rich in olive oil, vegetables, whole grains, and moderate protein intake.
  Interventions: Behavioral: Mediterranean diet

INTERVENTIONS:
Behavioral: Ketogenic diet — A structured, equicaloric ketogenic diet providing approximately 1200 kcal/day, consisting of high fat (70-80 g/day), moderate protein (80-90 g/day), and very low carbohydrate intake (20-30 g/day), primarily from non-starchy vegetables. The diet is administered for 3 consecutive weeks to induce nutritional ketosis. A sugar-free multivitamin supplement is provided throughout the intervention.
  Arms: Arm A - Ketogenic Diet (3 weeks)
Behavioral: Mediterranean diet — A structured Mediterranean diet administered for 3 weeks following a 2-week transition phase. The diet provides approximately 1200 kcal/day and emphasizes plant-based foods, extra virgin olive oil as the main fat source, moderate consumption of fish, dairy products, and whole grains, with limited red meat and processed foods.
  Arms: Arm B: Mediterranean Diet

SUMMARY:
This prospective, single-center, crossover study aims to evaluate the metabolic and hormonal effects of a ketogenic diet compared to a Mediterranean diet in patients with active acromegaly. Twenty-six adult patients with biochemically confirmed active acromegaly will undergo a three-week ketogenic diet followed by a three-week Mediterranean diet, with a two-week transitional phase. The primary outcome is the change in serum IGF-1 levels. Secondary outcomes include changes in anthropometric, biochemical, and inflammatory parameters. The study also explores the feasibility and safety of a structured ketogenic dietary intervention in this population.

DETAILED DESCRIPTION:
Acromegaly is a rare endocrine disorder characterized by excessive secretion of growth hormone (GH) and insulin-like growth factor 1 (IGF-1), often leading to metabolic complications including insulin resistance, diabetes mellitus, and hepatic steatosis. Nutritional status is a key regulator of the somatotropic axis, and recent evidence suggests that specific dietary patterns can modulate GH and IGF-1 secretion. The ketogenic diet (KD), characterized by high fat, moderate protein, and very low carbohydrate intake, induces nutritional ketosis, improves insulin sensitivity, and reduces circulating insulin levels. These effects may influence the hepatic expression of GH receptors and IGF-1 production. Preliminary data suggest that KD may reduce IGF-1 levels in patients with acromegaly.

This study is designed as a single-arm crossover trial involving 26 patients with active acromegaly. All participants will follow a structured ketogenic diet for three weeks (~1200 kcal/day, carbohydrates <30 g/day), followed by a two-week transition phase, and then a Mediterranean diet for three weeks (~1200 kcal/day, plant-based, rich in olive oil and fish). Baseline, post-KD, and post-Mediterranean assessments will include serum IGF-1 and GH levels, anthropometric measurements, body composition (via bioelectrical impedance analysis), liver enzymes, lipid profile, insulin resistance indices (HOMA-IR), and inflammatory markers (c-reactive protein, neutrophil to lymphocyte ratio, platelet to lymphocyte ratio).

The primary endpoint is the within-subject change in serum IGF-1 concentration. Secondary endpoints include changes in metabolic and inflammatory markers. Antidiabetic medications will be temporarily discontinued during the ketogenic phase under clinical supervision in patients not requiring insulin. The study is expected to provide novel insights into the impact of dietary modulation on the somatotropic axis in acromegaly and may inform future integrative therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of active acromegaly (elevated IGF-1, GH non-suppressible at OGTT)
* Stable medical therapy for ≥ 3 months
* BMI 25-40 kg/m²
* Informed consent signed

Exclusion Criteria:

* Type 1 diabetes or insulin-treated type 2 diabetes mellitus
* History of ketoacidosis
* Active malignancy, decompensated liver/kidney disease
* Severe psychiatric disorders or eating disorders
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Disease control | 3 weeks
  Change in serum IGF-1 levels after ketogenic and Mediterranean diets (paired comparison)

SECONDARY OUTCOMES:
Metabolic outcomes | 3 weeks
  Change in fasting glucose (mg/dL)
Metabolic outcomes | 3 weeks
  Change in fasting insulin (µU/mL)
Metabolic outcomes | 3 weeks
  Change in HOMA-IR (unitless)
Anthropometric outcomes | 3 weeks
  Change in body weight (kg)
Anthropometric outcomes | 3 weeks
  Change in Body Mass Index (BMI) (kg/m²)
Anthropometric outcomes | 3 weeks
  Change in waist circumference (cm)
Liver outcomes | 3 weeks
  Change in transaminases (U/L)
Lean and fat masses | 3 weeks
  Change in lean and fat mass (only after ketogenic diet)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This decision is based on institutional policy and ethical considerations, as the study involves a relatively small and identifiable patient population with a rare endocrine disorder. Data sharing may compromise patient confidentiality despite de-identification procedures.